CLINICAL TRIAL: NCT00376805
Title: Allogeneic Natural Killer Cells in Patients With Advanced Metastatic Breast Cancer
Brief Title: Allogeneic Natural Killer (NK) Cells in Patients With Advanced Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to toxicity
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMN-2005LS033; UMN-0505M70037 (Other: IRB, University of Minnesota); UMN-MT2005-08 (Other: Blood and Bone Marrow Transplantation Program); NCT00167193 (obsolete NCT alias)
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Results first posted 2010-08-12 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; male breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Whole-Body Irradiation; Radiation; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All Treated Patients (Experimental): All patients with advanced metastatic breast cancer treated with natural killer cells after receiving fludarabine, cyclosphosphamide and total body irradiation.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: Total body irradiation; Other: Natural killer cell infusion; Biological: Interleukin-2

INTERVENTIONS:
Drug: Fludarabine — administered intravenously 25 mg/m^2 times 5 doses
  Other Names: Fludara
Drug: Cyclophosphamide — administered intravenously 60 mg/kg days times 2 doses.
  Other Names: Endoxan, Cytoxan, Neosar, Procytox
Radiation: Total body irradiation — 200 cGy (gray) on day -1
  Other Names: radiation
Other: Natural killer cell infusion — Infused cell dose is within the range of 1.5-8.0 x 10^7/kg. Cell counts are based on total cells infused after the activation culture and washing determined on the morning of infusion.
  Other Names: NK cells
Biological: Interleukin-2 — administered subcutaneously (10 MU) 3 times per week for 6 doses
  Other Names: IL-2

SUMMARY:
RATIONALE: Giving chemotherapy before a donor natural killer (NK) cell infusion helps stop the growth of tumor cells. It also helps stop the patient's immune system from rejecting the donor's cells. Giving NK cells from a related donor may kill the tumor cells.

PURPOSE: This study furthers the research of previous studies (MT2003-01 and MT2004-25) which were to determine a specific preparatory regimen (cyclophosphamide and fludarabine) could create an environment in which infused NK cells can grow and effectively treat patients with relapsed AML. This study will test the previous regimen in patients with breast cancer.

DETAILED DESCRIPTION:
We believe that administration of related allogeneic (donor) natural killer cells along with IL-2, rather than autologous natural killer cells will provide the most effective anticancer therapy in this setting, and wish to test this approach. To do this, we will select a related donor who is partially HLA-matched with the study subject, to increase the likelihood that donor natural killer cells will kill the subject's cancer cells. We will also give chemotherapy drugs to increase the subject's tolerance for the donor natural killer cells. We will test the use of donor natural killer (NK) cell infusions. The immune system has a special way that it sees and identifies cancer cells or foreign agents (like viruses). The subject's own NK cells may not attack their cancer because NK cells see the tumor cells as "self" (a coating on the cell surface identifies a cell as "self" or "non-self"). We have reason to believe that NK cells may not kill cancer cells because NK cells have special receptors that "turn them off" when they encounter cancer cells (by seeing them as "self"). We may be able to get around this problem by using donor NK cells. Finally, subjects will receive a dose of subcutaneous IL-2 3 times a week (for 2 weeks) which has been proven safe in our previous studies to stimulate the natural killer cells.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of metastatic breast cancer that has progressed on or failed at least one salvage chemotherapy regimen for metastatic disease and that meets the following disease specific related criteria:

  * Measureable metastatic disease per Response Evaluation Criteria In Solid Tumor (RECIST) - bone only not eligible.
  * Disease progression while receiving prior therapy with a hormonal agent (if estrogen/progesterone receptor-positive) and/or trastuzumab (Herceptin®) (if HER2-neu positive)
  * Brain metastases allowed provided they are stable for ≥ 3 months after prior treatment
* Related HLA-haploidentical natural killer cell donor available (by ≥ class I serologic typing)
* Male or female
* Performance status 50-100%
* Platelet count ≥ 80,000/mm³ (unsupported by transfusions)
* Hemoglobin ≥ 9 g/dL (unsupported by transfusions)
* Absolute neutrophil count ≥ 1,000/mm³ (unsupported by sargramostim [GM-CSF] or filgrastim [G-CSF])
* Creatinine ≤ 2.0 mg/dL
* Liver function tests < 5 times normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* LVEF > 40%*
* Pulmonary function > 50%* (DLCO corrected AND FEV_1)
* No active infection (i.e., afebrile, off antibiotics, and no uninvestigated radiologic lesions)

Exclusion Criteria:

* At least 3 days since prior prednisone or other immunosuppressive medications
* No other concurrent therapy for cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-04; Primary Completion 2009-09 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Miller, MD, Study Chair — Masonic Cancer Center, University of Minnesota; Sarah Cooley, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- NK Cells With or Without Total Body Irradiation: Patients receiving natural killer cell infusion, fludarabine and cyclosphosphamide preparatory regimen, and with or without total body irradiation for treatment of metastatic breast cancer.
Period: Overall Study
Arm/Group | NK Cells With or Without Total Body Irradiation
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | NK Cells With or Without Total Body Irradiation
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Had Expansion of Natural Killer Cells
Description: Successful Natural Killer (NK) cell expansion is defined as detection of an absolute circulating donor-derived NK cell count of >100 cells/ul of whole blood 14 days after infusion with <5% donor T and B cells in mononuclear population (in metastatic breast cancer patients).
Time Frame: Day 14
Measure: Number; unit: Participants
Arm/Group | NK Cells With or Without Total Body Irradiation
Number analyzed (Participants) | 6
Participants | 0

2. Secondary Outcome: Number of Patients by Disease Response
Description: Defined by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria:
  * Complete Response (CR: Disappearance of all target lesions
  * Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR or sufficient increase to qualify for PD
  * Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions of appearance of one or more new lesions
  of clinical benefit (CB; stable disease for greater than 6 months.
Time Frame: 6 Months, 1 Year
Measure: Number; unit: Participants
Arm/Group | NK Cells With or Without Total Body Irradiation
Number analyzed (Participants) | 6
Participants
  Stable Disease | 4
  Progressive Disease | 2

3. Secondary Outcome: Number of Patients Who Died While on Study
Description: Number of patients who died within 100 days and after 100 days of natural killer (NK) treatment with or without total body irradiation.
Time Frame: Within 100 days, After 100 days
Measure: Number; unit: Participants
Arm/Group | NK Cells With or Without Total Body Irradiation
Number analyzed (Participants) | 6
Participants
  Died within 100 days | 1
  Died after 100 days | 5

4. Secondary Outcome: Overall Median Number of Days Patients Alive After Treatment
Description: Calculated median number of days of survival (patients alive days after treatment).
Time Frame: First Day of Treatment Until Death
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | NK Cells With or Without Total Body Irradiation
Number analyzed (Participants) | 6
Days | 124 [55 to 212]

ADVERSE EVENTS:
Time Frame: All adverse events were collected up to patients' death (within 1 year of treatment).
Arm/Group | NK Cells With or Without Total Body Irradiation
Serious Adverse Events (participants affected / at risk) | 6/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NK Cells With or Without Total Body Irradiation (N=6)
Bone marrow cellularity (Blood and lymphatic system disorders) | 1 (1) — Marrow aplasia
Death - disease progression NOS (General disorders) | 3 (3)
Death due to progressive disease (General disorders) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Passenger lymphocyte syndrome (Blood and lymphatic system disorders) | 1 (1) — Hemolysis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NK Cells With or Without Total Body Irradiation (N=6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (11)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (6)
Fever (General disorders) | 6 (26)
Chills (General disorders) | 6 (19)
Hypertension (Cardiac disorders) | 2 (12)
Hypotension (Cardiac disorders) | 1 (2)
Fatigue (General disorders) | 6 (46)
Edema (Blood and lymphatic system disorders) | 4 (22)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (15) — Includes pulmonary infiltrates
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 6 (26)
Rash (Skin and subcutaneous tissue disorders) | 5 (30) — Includes desquamation
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 4 (6)
Nausea (Gastrointestinal disorders) | 4 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (16) — Includes arthralgia
Sweats (Skin and subcutaneous tissue disorders) | 4 (16)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (10)
Anxiety (Nervous system disorders) | 1 (3)
Hematuria (Renal and urinary disorders) | 1 (1)
Cardiac function LVEF (Cardiac disorders) | 1 (3)
Hemolytic anemia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No